CLINICAL TRIAL: NCT02075775
Title: MOON Shoulder Instability-Cohort of Patients Undergoing Operative Treatment.
Acronym: MOONSI
Status: Recruiting | Type: Observational
Sponsor: Carolyn M Hettrich (Other)
Collaborators: University of Michigan (Other); University of California, San Francisco (Other); University of Kentucky (Other); Hospital for Special Surgery, New York (Other); University of Colorado, Denver (Other); Ohio State University (Other); Washington University School of Medicine (Other); Orthopedic Institute, Sioux Falls, SD (Other); Vanderbilt University (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor-Investigator, Carolyn M Hettrich, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201208835
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Other Instability, Shoulder; Dislocations; Subluxations; Recurrent Dislocation of Shoulder Region
Keywords: instability
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MOON Shoulder Instability: Patients indicated for Shoulder Instability surgery

SUMMARY:
This project will be a multi-center, prospective longitudinal cohort for all patients undergoing primary shoulder instability surgery, excluding isolated SLAP repairs. We will be looking for risk factors for recurrent instability, revision surgery, and poor outcomes. Patients will be asked to complete the RAND-36, ASES, Shoulder Activity, EQ-5D and WOSI outcome measures, as well as demographic and socioeconomic information. Surgeons will complete a form after surgery with information on radiographic findings, physical exam, surgical findings, and the repair. Patients will wear a sling post-operatively, and follow standardized rehabilitation protocols, including physical therapy.

Patients will be sent outcome questionnaires at 2, 6, 10, and 20 years after surgery.

DETAILED DESCRIPTION:
The objective of this prospective multicenter cohort study of patients undergoing surgery for glenohumeral instability is to identify the outcomes, and more importantly, the previously unknown predictors of sports function, activity level, general health, recurrent instability symptoms, and surgical failures following surgery. Patient information at the time of the surgery (demographics, validated outcome measures), in addition to the physical exam findings, shoulder pathology at the time of surgery, and surgical treatment will be obtained. The validated outcome instruments are American Shoulder and Elbow Surgeons Score, Western Ontario Shoulder Instability, Kerlan Jobe Overhand Athlete Score, Shoulder Activity Score, and RAND-36. Post-operative physical exam data will be obtained at 6 months after surgery. Patient reported outcomes will be repeated at 2, 6, 10, and 20 years post-operatively. Our multivariable analysis will identify which of the many factors related to the injury, intra-operative treatment, postoperative care, physical patient characteristics, and behavioral patient characteristics contribute to recurrence and poor outcome.

ELIGIBILITY:
Inclusion Criteria:

This is a prospective cohort study; there is no control group. Subjects that are included are all patients undergoing surgery for shoulder instability.

Inclusion criteria:

* Anterior, posterior, and inferior instability
* Ages 12-99
* Open and arthroscopic repair
* Revision of a previous shoulder instability repair
* Latarjet/bone augmentation

Exclusion Criteria:

* Workers compensation patients
* Prisoners
* Non-English speaker
* Not mentally competent
* Unable/unwilling to return for clinical follow-up
* Arthroplasty patients
* Rotator cuff tears
* Fractures

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential subjects are patients who are undergoing surgery of the labrum and/or capsule for shoulder instability
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2042-12 (Estimated)

PRIMARY OUTCOMES:
Predictors of worse patient outcomes (pain and/or reduced quality of life). | 2 years, 6 years, 10 years and 20 years
  Patients will fill out PRO's after surgery

SECONDARY OUTCOMES:
Predictors for recurrent instability | 2 years, 6 years, 10 years and 20 years
  Patients will be asked if they have had repeat surgery, recurrent dislocation, subluxation, as well as symptoms of instability on WOSI

OTHER OUTCOMES:
Predictors of shoulder osteoarthritis | 6 years, 10 years and 20 years
  Patients will fill out PRO's, symptomatic may return for xrays

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn M Hettrich, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Brian Wolf, MD, MS, Principal Investigator — University of Iowa
Locations (11):
- United States (11):
  - UCSF Orthopedic Institute, San Francisco, California
  - University of Colorado, Boulder, Colorado
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Ohio State University, Columbus, Ohio
  - Orthopedic Institute, Sioux Falls, South Dakota
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hettrich CM, Magnuson JA, Baumgarten KM, Brophy RH, Kattan M; MOON Shoulder Group; Bishop JY, Bollier MJ, Bravman JT, Cvetanovich GL, Dunn WR, Feeley BT, Frank RM, Kuhn JE, Lansdown DA, Benjamin Ma C, Marx RG, McCarty EC, Neviaser AS, Ortiz SF, Seidl AJ, Smith MV, Wright RW, Zhang AL, Cronin KJ, Wolf BR. Predictors of Bone Loss in Anterior Glenohumeral Instability. Am J Sports Med. 2023 Apr;51(5):1286-1294. doi: 10.1177/03635465231160286. Epub 2023 Mar 20. PMID 36939180
- [Derived] Brophy RH, Dunn WR; MOON Shoulder Group; Baumgarten KM, Bishop JY, Bollier MJ, Bravman JT, Feeley BT, Grant JA, Jones GL, Kuhn JE, Benjamin Ma C, Marx RG, McCarty EC, Ortiz SF, Smith MV, Wolf BR, Wright RW, Zhang AL, Hettrich CM. Factors Associated With Shoulder Activity Level at Time of Surgery and at 2-Year Follow-up in Patients Undergoing Shoulder Stabilization Surgery. Am J Sports Med. 2022 May;50(6):1503-1511. doi: 10.1177/03635465221085978. Epub 2022 Apr 20. PMID 35442106
- [Derived] Baron JE, Duchman KR, Hettrich CM, Glass NA, Ortiz SF; MOON Shoulder Group; Baumgarten KM, Bishop JY, Bollier MJ, Bravman JT, Brophy RH, Carpenter JE, Cox CL, Feeley BT, Frank RM, Grant JA, Jones GL, Kuhn JE, Lansdown DA, Benjamin Ma C, Marx RG, McCarty EC, Miller BS, Neviaser AS, Seidl AJ, Smith MV, Wright RW, Zhang AL, Wolf BR. Beach Chair Versus Lateral Decubitus Position: Differences in Suture Anchor Position and Number During Arthroscopic Anterior Shoulder Stabilization. Am J Sports Med. 2021 Jul;49(8):2020-2026. doi: 10.1177/03635465211013709. Epub 2021 May 21. PMID 34019439